CLINICAL TRIAL: NCT04571086
Title: 68-Ga-FAPI-PET for Tumor Detection: A Prospective Observational Trial
Brief Title: FAPI-PET for Tumor Detection
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, PD Dr. med. Wolfgang Fendler, MD, University Hospital, Essen
Other Study IDs: FAPI PET REG
Record Dates: First submitted 2020-09-15; First posted 2020-09-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Malignant Neoplasm
Keywords: FAPI; cancer; Positron-Emission-Tomography; FAP; fibroblast; imaging; PET
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood samples, tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational trial investigating correlation with histopathology, positive predictive value, detection rate, reproducibility and impact on clinical management of 68-Ga-FAPI PET/CT or PET/MRI in patients receiving this imaging modality for tumor staging or restaging as part of clinical care.

DETAILED DESCRIPTION:
68-Ga-fibroblast-activation-protein-inhibitors (68-Ga-FAPI) are novel Positron emission tomography (PET) tracers that were recently introduced for the imaging of patients with various cancer diseases. The fibroblast-activation-protein (FAP) is highly expressed in carcinoma-associated fibroblasts (CAFs) in the stroma of various tumor entities. The aim of this registry study is to collect data on FAPI expression, positive predictive value, detection rate, reproducibility and impact on clinical management of 68-Ga-FAPI PET/CT or PET/MRI on patients receiving this imaging modality at initial diagnosis or restaging as part of clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. FAPI-PET scheduled for staging or restaging as part of clinical routine for proven or suspected malignancy
2. Age ≥ 18 years.

Exclusion Criteria:

1. Patient cannot give consent for the study
2. Patient can not lie flat or tolerate FAPI PET imaging
3. Unwillingness or inability to comply with study and follow-up procedures
4. Condition of patient which is critical to participate in this study in the discretion of the investigators
5. Pregnant, lactating, or breast feeding women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for FAPI-PET for tumor staging or restaging
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between 68Ga-FAPI PET uptake intensity and histopathologic FAP expression. Validation via immunohistochemical FAP staining/molecular analyses of pathological specimen. | 3 Months

SECONDARY OUTCOMES:
Detection rate on a per-patient-basis of FAPI-PET for detection of tumor location, confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. | 3 Months
Detection rate on a per-region-basis of FAPI-PET for detection of tumor location, confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. | 3 Months
Positive predictive value (PPV) on a per-patient-basis of FAPI-PET for detection of tumor location, confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. | 3 Months
Positive predictive value (PPV) on a per-region-basis of FAPI-PET for detection of tumor location, confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. | 3 Months
Sensitivity and specificity of FAPI PET on a per-patient and per-region-basis for detection of tumor location confirmed by histopathology/biopsy (separate for regional, extra-regional and distant locations) | 3 Months
Impact on patient management assessed by pre- and post-imaging questionnaires | 12 Months
Detection rates on a per-patient basis of FAPI-PET stratified by tumor maker serum level and velocity | 12 Months
Rate of up- or downstaging following FAPI-PET imaging. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fendler, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- Department of Nuclear medicine, University hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watanabe M, Fendler WP, Grafe H, Hirmas N, Hamacher R, Lanzafame H, Pabst KM, Hautzel H, Aigner C, Kasper S, von Tresckow B, Stuschke M, Kummel S, Lugnier C, Hadaschik B, Grunwald V, Zarrad F, Kersting D, Siveke JT, Herrmann K, Weber M. Head-to-head comparison of 68 Ga-FAPI-46 PET/CT, 18F-FDG PET/CT, and contrast-enhanced CT for the detection of various tumors. Ann Nucl Med. 2025 Mar;39(3):255-265. doi: 10.1007/s12149-024-01993-7. Epub 2024 Oct 23. PMID 39443386